CLINICAL TRIAL: NCT01027546
Title: Effect of Tranexamic Acid on Reducing Postoperative Blood Loss in Cervical Laminoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yodakubo Hospital (Other)
Responsible Party: Takahiro Tsutsumimoto, Yodakubo hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YODA-0001
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2008-05

CONDITIONS: Cervical Myelopathy
Keywords: perioperative blood loss, spinal surgery
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- placebo, tranexamic acid (Placebo Comparator)
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Administer 15 mg/kg body weight of tranexamic Acid mixed in 100 mL saline intravenously over 15 min before the skin incision

SUMMARY:
The purpose is to evaluate the efficacy of tranexamic acid in cervical laminoplasty; the surgical procedure used was identical in all cases.

DETAILED DESCRIPTION:
Tranexamic acid, an inhibitor of fibrinolysis, has proven to be effective in reducing perioperative blood loss in patients undergoing total hip and knee arthroplasty. However, limited numbers of well-controlled trials in spinal surgery have been conducted due to heterogeneity in the performed surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled to undergo cervical laminoplasty from C3 to C6 for cervical multilevel compressive myelopathy with a narrow spinal canal for which nonoperative therapy had failed.

Exclusion Criteria:

* Patients with chronic renal failure, cirrhosis of the liver, serious cardiac disease, allergy to TXA, a history of thromboembolic disease, and bleeding disorders, as well as those who were currently receiving antiplatelet and/or anticoagulant drugs, were excluded from this study.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
perioperative blood loss | during and after surgery